CLINICAL TRIAL: NCT03496519
Title: A Phase I Study Assessing the Combination of Durvalumab (MEDI4736) and Trabectedin in Solid Tumors
Brief Title: Assessing the Combination of Durvalumab (MEDI4736) and Trabectedin in Solid Tumors
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Contract Issues
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 17-1852.cc
Record Dates: First submitted 2018-03-23; First posted 2018-04-12 (Actual); Last update posted 2018-10-09 (Actual); Status verified 2018-10

CONDITIONS: Solid Tumor, Adult
Keywords: Durvalumab; Trabectedin; Maximum Tolerated Dose; Lung Cancer; Sarcoma
MeSH Terms: conditions — Lung Neoplasms; Sarcoma | interventions — Trabectedin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Dose Escalation (Experimental): Dose escalation will occur following a 3+3 design in all advanced tumor types meeting the inclusion and exclusion criteria.
  * Cohort -1 (if necessary): Durvalumab 1125mg with Trabectedin 0.5mg/m2
  * Cohort 1: Durvalumab 1125mg with Trabectedin 0.75mg/m2
  * Cohort 2: Durvalumab 1125mg with Trabectedin 1.0mg/m2
  * Cohort 3: Durvalumab 1125mg with Trabectedin 1.2mg/m2
  * Cohort 4: Durvalumab 1125mg with Trabectedin 1.5mg/m2
  Interventions: Drug: Dose Escalation of Durvalumab and Trabectedin
- Dose Expansion (Experimental): Patients at this level will receive the safest dose of Durvalumab and Trabectedin that was determined during the Dose Escalation Phase. There will be a fixed dosage of Durvalumab, 1125mg, given intravenously over 60 minutes on Day 2 every 21 days. There will be fixed dosage of Trabectedin for each cohort, given through intravenous infusion as an outpatient, over a 24 hour period on Day 1 every 21 days.
  Interventions: Drug: Dose Expansion of Durvalumab and Trabectedin

INTERVENTIONS:
Drug: Dose Escalation of Durvalumab and Trabectedin — There will be a fixed dosage of Durvalumab, 1125mg, given intravenously over 60 minutes on Day 2 every 21 days. There will be an increase in Trabectedin for each cohort, given through intravenous infusion over a 24 hour period on Day 1 every 21 days as an outpatient.
  * Cohort -1: Durvalumab 1125mg with Trabectedin 0.5mg/m2
  * Cohort 1: Durvalumab 1125mg with Trabectedin 0.75mg/m2
  * Cohort 2: Durvalumab 1125mg with Trabectedin 1.0mg/m2
  * Cohort 3: Durvalumab 1125mg with Trabectedin 1.2mg/m2
  * Cohort 4: Durvalumab 1125mg with Trabectedin 1.5mg/m2
  Other Names: Combination of Durvalumab and Trabectedin
  Arms: Dose Escalation
Drug: Dose Expansion of Durvalumab and Trabectedin — There will be a fixed dosage of Durvalumab, 1125mg, given intravenously over 60 minutes on Day 2 every 21 days. There will be a fixed dosage of Trabectedin for each cohort, whatever was determined to be the safest dose during the Dose Escalation Phase, and it will be given through intravenous infusion over a 24 hour period on Day 1 every 21 days as an outpatient.
  Other Names: Combination of Durvalumab and Trabectedin
  Arms: Dose Expansion

SUMMARY:
A phase 1 study examining the combination of Durvalumab (MEDI4736) and Trabectedin in various solid tumor types. The study seeks to determine a safe dose of the combination of study drugs and then examine this dose in larger groups of patients of specific tumor types to evaluate its anti-tumor efficacy. Treatment will continue in patients who respond for up to 1 year.

DETAILED DESCRIPTION:
This study will include dose escalation and dose expansion phases.

In the dose escalation portion, patients with advanced cancer will be enrolled and treated with Durvalumab and Trabectedin. Durvalumab will be administered at the same dose in each dose escalation cohort, while the dose of Trabectedin will be progressively increased in different cohorts until the safest dose of the combination is determined.

In the dose expansion portion patients will be treated with the safest dose of the study drugs determined during the dose escalation phase. There will be two separate groups of patients treated at this dose to evaluate anti-tumor efficacy of the combination. One group will consist of non-small-cell lung cancer patients previously treated with PD-1 or PD-L1 inhibitors and another group will consist of an immunotherapy naive group of patients. This immunotherapy naive group of patients will include sarcoma and another tumor type, this other tumor type will be determined based on anti-tumor efficacy seen during the dose escalation.

The study drugs will be given intravenously every 3 weeks. Treatment will continue for up to one year or until disease progression.

ELIGIBILITY:
Inclusion Criteria at Screening and C1D1:

1. Ability to understand and the willingness to sign a written informed consent document
2. Written informed consent and any locally-required authorization (e.g., HIPAA in the USA) obtained from the patient prior to performing any protocol-related procedures, including screening evaluations
3. AGE ≥ 18
4. Alkaline phosphatase (ALP) level ≤ upper limit of normal (ULN)
5. Aspartate aminotransferase (AST) and alanine amino transferase (ALT) ≤ ULN
6. Bilirubin ≤ ULN, if total bilirubin is > ULN, measure direct/indirect bilirubin to evaluate for Gilbert's Syndrome (if direct bilirubin is within normal range, subject may be eligible)
7. Albumin ≥ 2.5 g/dL
8. CPK ≤ 2.5 xULN
9. Body weight > 30 kg
10. ECOG performance status 0-1
11. Evidence of post-menopausal status or negative urinary or serum pregnancy test for female pre-menopausal patients. Women will be considered post-menopausal if they have been amenorrheic for 12 months without an alternative medical cause. The following age-specific requirements apply:

    * Women <50 years of age would be considered post-menopausal if they have been amenorrheic for 12 months or more following cessation of exogenous hormonal treatments and if they have luteinizing hormone and follicle-stimulating hormone levels in the post-menopausal range for the institution or underwent surgical sterilization (bilateral oophorectomy or hysterectomy).
    * Women ≥50 years of age would be considered post-menopausal if they have been amenorrheic for 12 months or more following cessation of all exogenous hormonal treatments, had radiation-induced menopause with last menses >1 year ago, had chemotherapy-induced menopause with last menses >1 year ago, or underwent surgical sterilization (bilateral oophorectomy, bilateral salpingectomy or hysterectomy).
12. Evaluable disease for dose escalation, measurable disease per RECIST 1.1 for dose expansions
13. Hemoglobin ≥ 9 g/dL
14. Neutrophil count ≥ 1.5 x 10^9/L
15. Platelets ≥ 100 x 10^9/L
16. Measured creatinine clearance (CL) ≥ 50 mL/min or Calculated creatinine CL≥ 50 mL/min by the Cockcroft-Gault formula (Cockcroft and Gault 1976) or by 24-hour urine collection for determination of creatinine clearance:

    This calculation will be performed by a member of the clinical study team

    Males:

    Creatinine CL (mL/min) = Weight (kg) x (140 - Age) / 72 x serum creatinine (mg/dL)

    Females:

    Creatinine CL (mL/min) = [Weight (kg) x (140 - Age)/72 x serum creatinine (mg/dL)] x 0.85
17. Any advanced unresectable/stage IV solid tumor with exception of primary CNS malignancy is permitted.
18. Enrolled patients may be candidates for standard of care therapy with trabectedin or second line/subsequent line treatment for advanced disease with PD-1/PD-L1 inhibitor monotherapy. Otherwise they should have no standard of care option available or be felt appropriate for a phase I clinical trial in the opinion of the treating investigator. Prior PD-1/PD-L1 exposure is not an exclusion criteria.
19. For the expansion cohort of NSCLC patients previously treated with and having progressed on immunotherapy patients must have no standard of care option available or have contraindications to such treatment (including those who decline such treatment).
20. Patient is willing and able to comply with the protocol for the duration of the study including undergoing treatment and scheduled visits and exams including follow up.

Exclusion Criteria:

1. Strong inhibitors or inducers of cytochrome P450 3A (washout from prior use of such agents before C1D1 must exceed 21 days).
2. Concurrent enrollment in another clinical study, unless it is an observational (non-interventional) clinical study or during the follow-up period of an interventional study.
3. Receipt of the last dose of anticancer therapy (chemotherapy, immunotherapy, endocrine therapy, targeted therapy, biologic therapy, tumor embolization, monoclonal antibodies or other investigational product) ≤ 28 days. However, if a therapy has a short half-life, then patients may participate if they received prior treatment ≤ 28 days before starting study treatment with approval from the PI and AstraZeneca/Janssen. Acceptable washout periods include:

   1. 3-14 days for prior TKI depending on half-life
   2. 14-28 days for prior PD-1 or PD-L1 inhibitor treatment depending on the frequency of administration (i.e., wait one full cycle of prior PD-1 axis inhibition before starting study drugs)
4. Therapeutic radiation within 6 weeks of cycle 1 day 1. Exceptions are palliative radiation and/or stereotactic radiation to non-target lesions.
5. If received prior immunotherapy must not have experienced one of the following:

   * A toxicity that led to permanent discontinuation of prior immunotherapy
   * All AEs while receiving prior immunotherapy must have completely resolved or resolved to baseline prior to screening for this study.
   * Must not have experienced a ≥Grade 3 immune related AE or an immune related neurologic or ocular AE of any grade while receiving prior immunotherapy. NOTE: Patients with endocrine AE of ≤Grade 2 are permitted to enroll if they are stably maintained on appropriate replacement therapy and are asymptomatic.
   * Must not have required the use of additional immunosuppression other than corticosteroids for the management of an AE and must not have experienced recurrence of an AE if re-challenged.
6. Prior treatment with trabectedin or trabectedin analog
7. History of another malignancy except for:

   * Malignancy treated with curative intent and with no known active disease ≥5 years before the first dose of study drugs and of low potential risk for recurrence
   * Adequately treated non-melanoma skin cancer or lentigo maligna without evidence of disease
   * Adequately treated carcinoma in situ without evidence of disease e.g., cervical cancer in situ
8. Mean QT interval corrected for heart rate (QTc) > 450 ms for males or > 470 msec for females calculated from 3 electrocardiograms (ECGs) using Fredericia's Formula (within at least 15 minutes, at least 5 minutes apart)
9. Current or prior use of systemic immunosuppressive medication within 28 days before the first dose of durvalumab + trabectedin, with the exception of systemic corticosteroids at physiological doses, which are not to exceed 10 mg/day of prednisone, or an equivalent corticosteroid. The following are exceptions to this criterion:

   - Steroids as premedication for hypersensitivity reactions (e.g., CT scan premedication)
10. Any unresolved toxicity (non-immune mediated) NCI CTCAE Grade ≥ 2 from previous anticancer therapy with the exception of alopecia

    - However, patients with irreversible toxicity not reasonably expected to be exacerbated by the treatment with durvalumab + trabectedin may be included only after consultation with the Principal Investigator.
11. Major surgical procedure (as defined by the Investigator) within 28 days prior to the first dose of study drugs. Note: Local surgery of isolated lesions for palliative intent is acceptable.
12. History of allogenic organ transplantation (both solid organ and bone marrow)
13. Active or prior documented autoimmune or inflammatory disorders (including inflammatory bowel disease [e.g., colitis or Crohn's disease], diverticulitis [with the exception of diverticulosis], systemic lupus erythematosus, Sarcoidosis syndrome, or Wegener syndrome [granulomatosis with polyangiitis, Graves' disease, rheumatoid arthritis, hypophysitis, uveitis, etc]). The following are exceptions to this criterion:

    * Patients with vitiligo or alopecia
    * Patients with hypothyroidism (e.g., following Hashimoto syndrome) stable on hormone replacement
    * Any chronic skin condition that does not require systemic therapy
    * Patients without active disease in the last 5 years may be included, but only after consultation with the PI
    * Patients with celiac disease controlled by diet alone
14. Uncontrolled intercurrent illness, including but not limited to, ongoing or active infection, symptomatic congestive heart failure, uncontrolled hypertension, unstable angina pectoris, cardiac arrhythmia, interstitial lung disease, serious chronic gastrointestinal conditions associated with diarrhea, or psychiatric illness/social situations that would limit compliance with study requirements, substantially increase risk of incurring AEs or compromise the ability of the patient to give written informed consent.
15. Cirrhosis of any Child Pugh class
16. Left ventricular ejection fraction less than 50%
17. History of pulmonary fibrosis, organizing pneumonia, drug-induced pneumonitis, idiopathic pneumonitis or evidence of symptomatic interstitial lung disease on chest computed tomography (CT).
18. History of leptomeningeal carcinomatosis
19. Has untreated central nervous system (CNS) metastases and/or carcinomatous meningitis that meets RECIST criteria identified either on the baseline brain imaging obtained during the screening period or identified prior to signing the informed consent form (ICF). Patients whose brain metastases have been treated may participate provided they show radiographic stability (defined as 2 brain images, both of which are obtained after treatment to the brain metastases. These imaging scans should both be obtained at least four weeks apart and show no evidence of intracranial progression). In addition, any neurologic symptoms that developed either as a result of the brain metastases or their treatment must have resolved or be stable either, without the use of steroids, or are stable on a steroid dose of ≤10mg/day of prednisone or its equivalent and not requiring anticonvulsants for at least 14 days prior to the start of treatment.
20. History of active primary immunodeficiency
21. Active infection including tuberculosis (clinical evaluation that includes clinical history, physical examination and radiographic findings, and TB testing in line with local practice), hepatitis B (HBsAg positive), hepatitis C, or human immunodeficiency virus (positive HIV 1/2 antibodies). Patients with a past or resolved HBV infection (defined as the presence of hepatitis B core antibody [anti-HBc] and absence of HbsAg) are eligible. Patients positive for hepatitis C (HCV) antibody are eligible only if polymerase chain reaction is negative for HCV RNA.
22. Receipt of live attenuated vaccine within 30 days prior to the first dose of study drugs. Note: Patients, if enrolled, should not receive live vaccine whilst receiving treatment with study drugs and up to 90 days after the last dose of study drugs.
23. Female patients who are pregnant or breastfeeding or male or female patients of reproductive potential who are not willing to employ effective birth control (as defined in section 7.1 of protocol) from screening to 180 days after receipt of the last dose of study drugs.
24. Known allergy or hypersensitivity to any of the study drugs or any of the study drug excipients.
25. Prior randomisation or treatment in a previous durvalumab and/or tremelimumab clinical study regardless of treatment arm assignment.
26. Judgment by the investigator that the patient is unsuitable to participate in the study and the patient is unlikely to comply with study procedures, restrictions and requirements.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-10-01 (Estimated); Primary Completion 2021-10-31 (Estimated); Study Completion 2021-10-31 (Estimated)

PRIMARY OUTCOMES:
Recommended Dosage of the Durvalumab and Trabectedin Combination | Up to 1 year on study treatment plus 90 days safety follow-up, up to 15 months
  Recommended Phase II Dose (RP2D) is the dose determined safest for further evaluation based on both early and late onset side effects detected during the dose escalation phase.
Maximum tolerated dose | First 2 cycles at 21 days each, equal to 42 days.
  Maximum Tolerated Dose (MTD) is defined as the highest dose level with no more than 1 Dose Limiting Toxicity (DLT) reported out of up to 6 DLT-evaluable subjects determined during the dose escalation phase

SECONDARY OUTCOMES:
Overall Response Rate (ORR) of the Durvalumab and Trabectedin Combination in the whole treated population and at the RP2D in the expansion cohort(s) | After 2 cycles of study drugs to study end date, up to 24 months.
  ORR is determined by RECIST v1.1 and iRECIST response criteria.
Duration of Response (DOR) of the Durvalumab and Trabectedin Combination | After 2 cycles of study drugs, up to 24 months.
  The time period for which a partial response (PR) or complete response (CR) is maintained.
Clinical Benefit Rate (CBR) of the Durvalumab and Trabectedin Combination | After 2 cycles of study drugs to study end date, up to 24 months.
  Determined by complete response, partial response, or stable disease.
One Year Progression Free Survival (PFS) of the Durvalumab and Trabectedin Combination | Study start date to progression, or death, whichever comes first, up to 24 months.
  PFS is determined by RECIST v1.1 and iRECIST
One Year Overall Survival (OS) of the Durvalumab and Trabectedin Combination | Study start date to death from any cause, up to 24 months.
  Determined continuously throughout the study.
Incidence of Treatment-Emergent Adverse Events (Safety) | Study start date to study end date, up to 24 months.
  Number of participants with abnormal laboratory values and/or adverse events that are related to treatment.
Incidence of Treatment-Emergent Adverse Events (Tolerability) | Study start date to study end date, up to 24 months.
  Number of participants with abnormal laboratory values and/or adverse events that are related to treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Jose Pacheco, Principal Investigator — University of Colorado, Denver